CLINICAL TRIAL: NCT06485882
Title: Examining the Effectiveness of Education Based on Social Learning Theory in Fostering Self-care and Social Skills in School Children: A Randomized Controlled Trial
Brief Title: Examining the Effectiveness of Education Based on Social Learning Theory in Fostering Self-care and Social Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Isın Alkan, Research Assistant Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 'HacettepeU'
Record Dates: First submitted 2024-04-05; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Main Heading (Descriptor) Terms
Keywords: Social learning theory; Self-care; Social competence; Preschool period
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Intervention Model Description: Social Learning Theory is used for fostering positive health habits for children between 5-6 age.
Who Masked: Care Provider
Masking Description: Teachers fullfilled the scales and so they were not known about children who are intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention Group Procedure Children in the intervention group, who met the inclusion criteria for the study and agreed to participate, were informed about the training they were to receive. Teachers were also informed about the self-care and social competence scales they were to administer to the children.
  Interventions: Behavioral: Self-Care Training
- Control group (No Intervention): The self-care and social competence skills of the children in the control group were assessed at the beginning of the study together with the intervention group. To this end, pretests of the Self-Care Skills Assessment Scale for 3- to 6-Year-Old Children, and the Social Competence and Behavior Evaluation - 30 Scale were filled out by the teachers, while the parents were asked to fill out the Demographic Assessment Form.
  Posttest: The children in the control group received no extra self-care or social competence training besides that provided by the teachers for one week as part of the regular curriculum. For the posttest of this group, the Self-Care Skills Assessment Scale for 3- to 6-Year-Old Children was used, as well as the Social Competence and Behavior Evaluation-30 Scale, both of which were filled out by the teachers at the end of the fourth month. No other assessments were carried out in the intervening months.

INTERVENTIONS:
Behavioral: Self-Care Training — Animation films are watched children about self-care and social competence
  Other Names: Social Competence Training
  Arms: Intervention group

SUMMARY:
Abstract Purpose: This study was conducted to examine the effectiveness of a training program prepared on the basis of the Social Learning Theory for teaching self-care and social competence behaviors in preschool children.

Design and method: The sample of the study consisted of 41 in the intervention and 41 in the control group. Data were collected using the Demographic Assessment Form, the Self-Care Skills Assessment Scale and the Social Competence and Behavior Evaluation-30 Scale. Using five animated films created on the basis of the Social Learning Theory for fostering children self-care and social competence behaviors, a total of 20 training sessions were conducted with intervention group over a period of four months. Self-care and social competence scales were administered at the end of each month. Ultimately, children were assessed a total of five times.

DETAILED DESCRIPTION:
Preschool is a period in the life of children when they experience rapid cognitive and social development, and their capacity for learning is at its greatest. In this period, children have a natural curiosity and a desire to learn everything they can, make observations and duplicate the behaviors of others.

Preschool is an important time of life when behaviors are shaped, habits are formed and basic health-related behaviors are acquired, with self-care being one of the most important acquired behaviors in this period for personal health. Self-care skills can be defined as the daily life skills required for a child to be able to meet their basic needs on their own, without the help of an adult, at home, at school or in other settings. The self-care skills that children acquire as they develop, such as those related to eating, dressing, personal care and toileting, are vital components of a bio-psycho-socially healthy life. Self-care plays an important role in the development of positive health behaviors and quality of life.

The healthy self-care behaviors expected from preschool children include an ability to wash oneself without wetting one's clothes, brushing teeth at least twice a day without help, toilet hygiene, healthy eating and nutritional habits, dressing skills, separating clean and dirty clothes, dressing for the weather, covering one's mouth when sneezing or coughing, using a tissue to wipe a runny nose and combing one' hair without help. Social learning refers to learning in a social environment. Social learning theory argues that human behaviors are shaped by the interactions between cognitive, behavioral and environmental factors. According to social learning theory, learning takes place via reactions and modeling. Bandura, a leading proponent of social learning theory, claims that many behaviors are learned through the observation and modeling of the behaviors of others.

Positive peer relationships in preschool help children adapt to school and acquire emotional control, conflict resolution and self-regulation skills, while also improving their social competencies, and contributing to their psychosocial, cognitive, affective and moral development. In this period, peers function as sources of information, models and interlocutors, and facilitate the learning of new knowledge, skills and behaviors.

Contemporary media, including smartphones, tablets, PCs and television, in particular, play an undeniable role in observation- and modeling-based learning among children. Children have at their disposal a wealth of technological devices through which they can interact with others at all hours of the day, providing them with easy access to information and other content that can shape their individual behaviors. The important role played by the media in social learning should not be underestimated.

Social learning theory is based on the fact that children identify with characters in TV shows, and cartoons in particular, and adopt the behaviors and attitudes displayed by those characters by making a conscious effort to copy them. Cartoon characters on TV play an important role both in shaping the characters of children, and can aid them in the acquisition of health-related behaviors.

In order to create a healthy society in the future, the training to be given to children in the preschool period about self-care and social competence and the methods to be used in this training are of critical importance. There is, however, a need for effective intervention programs targeting the improvement of self-care skills and social competence levels in children. Given the long-term negative effects of deficiencies in social competence and emotional control skills, it is of great importance for school nurses to identify at-risk children as early as possible and provide guidance for proper counseling. It is very important for nurses to implement health-promoting nursing interventions in order to ensure that the child is best prepared for life and has the chance to realize himself throughout his life. School nurses can thus play an important role in training parents and preschool teachers on the acquisition of positive health behaviors by children.

A review of literature revealed a lack of training programs in Türkiye that use animated cartoon characters to improve the self-care and social competence skills of children. This research was conducted to examine the effectiveness of a training program based on social learning theory in teaching self-care (general body hygiene, nose and ear cleaning, dental health, hand hygiene) and social competence skills to children five and six years of age. The hypotheses tested in the study are presented in the following.

Hypotheses Hypothesis 1. Following the training based on social learning theory, the intervention group differs from the control group in terms of self-care behaviors.

Hypothesis 2. Following the training based on social learning theory, the intervention group differs from the control group in terms of social competence skills.

Methods Design and Sample A randomized controlled intervention design was used in this study. The population of the study consisted of official kindergartens affiliated with the Ministry of National Education in a province. The selected province had 25 districts, one of which was selected using simple random sampling. This district had 18 official kindergartens affiliated with the Ministry of National Education, and one was selected using simple random sampling.

Participants and randomization

The power analysis conducted using the software G*Power 3.0.10 showed that in a study design with 5 repetitions and 2 groups (intervention and control), a sample size of 82 was required for an effect size of 0.7362, power of 95% power, and 5% margin of error. The two kindergartens included in the study had a total of 180 children five and six years of age. A list of these children was created, each child was given a number, and lots were drawn from a box containing pieces of paper with these numbers on them. The first number drawn was assigned to the intervention group, the second number to the control group, and so on, until the intervention and control group had 43 participants each. Thus, given the risk of attrition, a total of 86 children were included in the study, all of whom were five or six years of age, agreed to participate in the study, and had parents who gave their written consent for the study (Figure 1 CONSORT).

To test the comprehensibility of the cartoons prepared and the data collection forms, a pilot study was conducted with 10 children attending one of the schools sampled. G*Power analysis was based on data from this pilot study. Children who participated in the pilot study were excluded from the main study.

Blinding It was not possible to blind the researchers to the intervention and control groups for randomization. However, the data collection process was blinded by using classroom teachers who work in the kindergarten included in the study. Self -care and social competence scales were administered by the teachers who were unaware of the intervention and control groups of the children.

Variables Mean scores of the intervention and control groups on the self-care, social competence and behavior evaluation scales were the dependent variables. Independent variables were the training program -which involved animated films on self-care and social competence skills- and sociodemographic variables.

Intervention Group Procedure Pretest: In this session, children in the intervention group, who met the inclusion criteria for the study and agreed to participate, were informed about the training they were to receive. Teachers were also informed about the self-care and social competence scales they were to administer to the children.

To have pretest measurements prior to the training program, the Self-Care Skills Assessment Scale and the Social Competence and Behavior Evaluation-30 Scale were distributed to the teachers to be filled out, while the parents were asked to fill out the Demographic Assessment Form.

ELIGIBILITY:
Inclusion Criteria:

* Children who were five or six years of age and did not have any cognitive or sensory issues were included in the study.

Exclusion Criteria:

* Children with cognitive or sensory issues requiring special education were not included in the study.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Fostering self-care behaviours | The study lasted 30 weeks in totally
  Total of 20 training sessions were organized over four months based on the stages defined in the Social Learning Theory, and animated films focusing on target behaviors related to self-care was used as training tools. For evaluating the changes of behaviors the Self-Care Skills Assessment Scale was used. Positive changes were observed in the self-care behaviors of the children after the implemented education program. The total score of the self-care scale increased more in the intervention group than in the control group. The minimum score that the children received from Scale was calculated as 205, and the maximum score was 241. It was reported whether there was a change in children's self-care behaviors with the analyses made. The Self-Care Skills Assessment Scale used in these measurements was applied separately for each case.
Fostering social skills in school children | At the end of the monthly training sessions for the intervention group, evaluations were made with scales every month, and it lasted 30 weeks in totally.
  Total of 20 training sessions were organized over four months based on the stages defined in the Social Learning Theory, and animated films focusing on target behaviors related to social competence was used as training tools. For evaluating the changes of behaviors the Social Competence and Behavior Evaluation-30 Scale was used. Positive changes were observed in the social competence behaviors of the children after the implemented education program. The total score of the social competence increased more in the intervention group than in the control group. The minimum score that the children received from Scale was calculated as 44, and the maximum score was 54. It was reported whether there was a change in children's social competence behaviors with the analyses made. The the Social Competence and Behavior Evaluation-30 Scale used in these measurements was applied separately for each case.

SECONDARY OUTCOMES:
Hygiene and self care | The study lasted 30 weeks in totally
  Total of 20 training sessions were organized over four months based on the stages defined in the Social Learning Theory, and animated films focusing on target behaviors related to hygiene and personal care was used as training tools. For evaluating the changes of behaviors the Self-Care Skills Assessment Scale was used. Positive changes were observed in the hygiene and personal care behaviors of the children after the implemented education program. The total score of the hygiene and personal care increased more in the intervention group than in the control group. The minimum score that the children received from The Self-Care Skills Assessment Scale was calculated as 79, and the maximum score was 90. It was reported whether there was a change in children's hygiene and personal care behaviors with the analyses made. The Self-Care Skills Assessment Scale used in these measurements was applied separately for each case.

OTHER OUTCOMES:
Anger-Aggression | The study lasted 30 weeks in totally.
  Total of 20 training sessions were organized over four months based on the stages defined in the Social Learning Theory, and animated films focusing on target behaviors related to anger-agression was used as training tools. For evaluating the changes of behaviors the Social Competence and Behavior Evaluation-30 Scale was used. Positive changes were observed in the anger-agression behaviors of the children after the implemented education program. The total score of the anger-agression decreased more in the intervention group than in the control group. The minimum score that the children received from The Social Competence and Behavior Evaluation-30 Scale was calculated as 10, and the maximum score was 16. It was reported whether there was a change in children's Social Competence and Behavior Evaluation-30 Scale behaviors with the analyses made. The Social Competence and Behavior Evaluation-30 Scale used in these measurements was applied separately for each case.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denham SA, Bassett HH, Way E, Mincic M, Zinsser K, Graling K. Preschoolers' emotion knowledge: self-regulatory foundations, and predictions of early school success. Cogn Emot. 2012;26(4):667-79. doi: 10.1080/02699931.2011.602049. Epub 2011 Aug 19. PMID 21851307
- [Background] Ghasemi A, Zahediasl S. Normality tests for statistical analysis: a guide for non-statisticians. Int J Endocrinol Metab. 2012 Spring;10(2):486-9. doi: 10.5812/ijem.3505. Epub 2012 Apr 20. PMID 23843808
- [Background] Guhn, M., Gadermann, A.M., Almas, A., Schonert-Reichl, K.A., & Hertzman, C. (2016). Associations of teacher-rated social, emotional, and cognitive development in kindergarten to self-reported wellbeing, peer relations, and academic test scores in middle childhood. Early Childhood Research Quarterly, 35, 76-84. doi: 10.1016/j.ecresq.2015.12.027.
- [Background] Halford JC, Boyland EJ. The marketing of foods and non-alcoholic beverages to children. Setting the research agenda. Appetite. 2013 Mar;62:182-4. doi: 10.1016/j.appet.2012.12.003. Epub 2012 Dec 7. No abstract available. PMID 23220356
- [Background] Jones, S.M., McGarrah, M.V., & Kahn, J. (2019). Social and emotional learning: A principled science of human development in context. Educational Psychologist, 54(3), 129-143.
- [Background] Koh, K.L., & Ahad, N.A. (2020). Normality for non-normal distributions. Journal of Science and Mathematics Letters, 8(2), 51-60.
- [Background] Rai, S., Waskel, B., Sakalle, S., Dixit, S., & Mahore, R. (2016). Effects of cartoon programs on behavioural, habitual and communicative changes in children. International Journal of Community Medical Public Health, 3, 1375-1378.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT06485882/Prot_SAP_ICF_000.pdf